CLINICAL TRIAL: NCT05375500
Title: Embodiment in Virtual Reality as a Telemedicine Digital Therapeutic for the Treatment of Chronic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karuna Labs Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2022-03-28; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain; Low Back Pain; Shoulder Pain
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Digital Therapeutic Arm (Experimental): measure the treatment effects of digital therapeutic intervention
  Interventions: Device: telemedicine digital therapeutic

INTERVENTIONS:
Device: telemedicine digital therapeutic — digital therapeutics intervention for chronic pain utilizing coaching and virtual reality application

SUMMARY:
Chronic shoulder pain is a common musculoskeletal pain condition that can have a profound impact on a sufferer's life and a large socioeconomic healthcare burden to society. The aim of this study was to determine the feasibility of delivering telemedicine enabled functional shoulder rehabilitation for chronic shoulder pain patients using immersive virtual reality. Ten chronic shoulder pain patients were recruited from local pain clinics. Patients engaged in three sessions of virtual embodiment training per week over the course of eight weeks. Rehabilitation sessions were delivered on an Oculus Quest head-mounted display and hand controllers. Rehabilitation exercises (virtual embodiment training) leverage techniques from graded motor imagery, such as visual mirror feedback and augmentation of the virtual avatar's movements. Eight pain assessments were administered prior to the first session, and at weeks four and eight to get an indication of the effect that telemedicine delivered virtual embodiment training has on symptoms of chronic shoulder pain.

DETAILED DESCRIPTION:
This study protocol was conducted in accordance with the ethical standards of the Declaration of Helsinki and approved by ADVARRA, an independent institutional review board. Ten chronic shoulder pain patients (7 Female, 3 Male, mean age = 48.44 years) provided written informed consent prior to participating in the study. Eight patients presented with chronic pain of the left shoulder and two presented with right chronic shoulder pain. Patients were recruited from a local pain clinic. Patients were excluded if they reported a history of motion sickness, a history of seizures, or cognitive impairments. A total of twenty-one patients were assessed for eligibility. Two patients were excluded prior to participation for a history of vertigo or motion sickness, and one was excluded due to color blindness. Four patients declined to participate prior to beginning treatment. Four patients were excluded due to impending surgeries scheduled that would prevent them from completing the study protocol (see Figure 1 consort diagram).

Patients who volunteered to participate in the study were shipped an Oculus Quest six-degrees-of-freedom wireless head mounted VR display (HMD) and hand controllers. Patients were assigned a health coach to assist with the use of the VR hardware. The health coach met with the patients via a HIPAA compliant telehealth video chat platform. Patients were instructed on safe use of the VR headset and hand controllers and instructed on how to create the safe play guardian of the Oculus Quest VR system and how to connect the HMD to a home wi-fi. After the patients confirmed that they were comfortable using the Oculus Quest, they were advised to complete three sessions of functional rehabilitation in VR exercises per week over the course of eight weeks. All function rehabilitation exercises were self-administered by each patient. The coach conducted telehealth video chat sessions with each patient once per week and administered a structured curriculum that included pain neuroscience education, goal setting, instructions for pacing and grading, and flare-up management.

Functional rehabilitation exercises were delivered through KarunaHOME (Karuna Labs, Inc, San Francisco, CA). KarunaHOME is a virtual reality software delivered on the oculus quest to provide rehabilitation exercises in patient's homes. KarunaHOME Virtual Embodiment Training™ consists of five functional rehabilitation exercises designed on the principles of graded exposure and mirror therapy.

Each session of functional rehabilitation began with a calibration exercise that measured shoulder range of motion for flexion, scaption, and abduction (Figure 2). The calibration exercise progressed through shoulder flexion, shoulder scaption, and shoulder abduction one at a time, on each side. The patient was instructed in VR to perform three repetitions within a comfortable range. The calibration exercise was a measurement of a patient's comfortable range of motion for flexion, scaption, and abduction and was used to set the limits of subsequent exercises so that patient did not move beyond their comfortable range during that day's session. The second exercise was a functional movement exercise that promoted shoulder flexion, scaption, and abduction while engaged in a reach and grasp task. Patients reached for an orb in the form of a floating lotus flower positioned in front of the patient in the virtual environment. Patients grasped the orb by moving the hand controller, which corresponded to movement of the virtual avatar's arm, and then pulled the trigger of the Oculus Quest hand controller using the index finger to toss the orb into a pond by producing either an overhand or underhand throwing motion and releasing the trigger. The second exercise also incorporated a mirror visual feedback (MVF) manipulation where the avatar's contralateral limb moved relative to the patient's movement. For example, if the patient moved their right arm, they would see embodied avatar's left arm moving. MVF was used for half the duration of each exercise. The third exercise was a reach and grasp exercise where patients reached to grasp colorful flowers by moving the hand controller to position the virtual avatar's arm in front of their embodied virtual avatar. The goal of this exercise was to match flowers of the same color in sets of three or more. The patient reached up for a flower to remove it and then the flowers above will fall into place. The exercise required patients to reach a maximum height by continuing to remove flowers. The fourth exercise was a painting exercise designed to promote complex dynamic shoulder motion. The goal of this exercise was to connect numbered dots by using the hand controller to move the virtual avatar's arm in a dynamic pattern to recreate different shapes in the sky using a virtual paintbrush. The first few shapes were directly in front of the patient and were simple movements such as a circle, triangle, heart. The shapes became progressively more difficult, requiring greater shoulder range of motion for reaching above and to the side, and progressed to more complex shapes to connect. The final exercise was a simulated activity of daily living in the form of a bow and arrow experience. Movements were designed to mimic motions that are included in activities of daily living such as putting on a seatbelt or shampooing hair. There were three distinct exercises within the bow and arrow activity. In all exercises, the patient moved the hand controller to move the virtual avatar's upper extremity limbs in a position that was necessary to complete the task. The first exercise required patients to reach the affected arm across body (horizontal adduction) to the quiver on the opposite hip to grasp an arrow and then bring the arrow to the bow (shoulder flexion) and pull back (scapular retraction) and shoot towards a target. The second exercise required patients to reach with affected arm over and behind the opposite shoulder to the quiver to get an arrow and then bring the arrow to the bow (shoulder flexion) and pull back (scapular retraction) and shoot. The third exercise required patients to reach over the affected shoulder (shoulder flexion, abduction, and internal and external rotation). Each session progressed from the first exercise to the last exercise with one minute of a guided breathing exercise in between each exercise. Patients completed three sessions per week over the course of eight weeks.

Telehealth-based pain education and behavioral health coaching was administered once per week. The first session was ninety minutes in duration and consisted of a general introduction, a tutorial on safely using the VR hardware in the home, and general introductions to Virtual Embodiment Training. Sessions two through eight were sixty minutes in duration with each session addressing topics that could be applied in the virtual embodiment exercises as well as activities of daily living. Each session included discussions of goals to work towards, including goals within virtual embodiment exercises. Sessions also contained pain neuroscience education, instruction on graded exposure, and behavioral exercises designed to help patients cope with their chronic pain and manage stress with relaxation, awareness of emotions and pain-related thoughts, mindfulness and gratitude-based exercises.Patients were encouraged to apply what they learned in the behavioral coaching sessions in exercised performed in VR.

The primary objective of this study was to assess the feasibility of a home-based functional rehabilitation program delivered in VR combined with telehealth-based education and coaching. The secondary objective was to determine appropriate outcome measures for an eventual larger scale randomized controlled trial. To assess the potential effectiveness of VR telehealth delivered functional rehabilitation, a battery of pain assessments were administered at three timepoints (pre, mid, and post), prior to beginning the eight week protocol, at the midpoint (week 4), and after completing the eight week protocol. The Disability of the Arm, Shoulder, and Hand (DASH) questionnaire was used to assess shoulder disability. The SF-36 was used to assess was administered to assess quality of life. The Pain Catastrophizing Scale (PCS) was used to assess psychological aspects of pain. The Fear Avoidance Beliefs Questionnaire (FABQ) physical activity subscale was used to assess fear of movement due to chronic pain. The Upper Extremity Functional Index (UEFI) was used to assess shoulder function. The Tampa Scale of Kinesiophobia (TSK) was used to assess fear of movement. The Pain Self-Efficacy Questionnaire (PSEQ) was used to assess patient confidence. The Yellow Flag Risk Form (YFRF) was used to assess chronic pain mechanisms. Since this was a feasibility study, additional measures were assessed to determine appropriate outcome measures for an eventual larger randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to wear a VR HMD (head-mounted display)
* Able to attend visits with the frequency outlined in the protocol

Exclusion Criteria:

* Individuals who have a cognitive impairment
* Susceptibility to motion sickness or simulator-sickness
* History of susceptibility to seizures per subject's reporting
* Pain due to skin infections
* Pain due to blood clots

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand | 1-2 months
  30-item questionnaire that evaluates disability performing upper extremity activities. This questionnaire is a self- report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale.
Upper Extremity Functional Index | 1-2 months
  The Upper Extremity Functional Index (UEFI) is a patient reported outcome measure used to assess the functional impairment in individuals with musculoskeletal upper limb dysfunction. The original UEFI consists of 20 questions on a 5- point rating scale assessing level of difficulty in performing activities of daily living using the upper extremities including household and work activities, hobbies, lifting a bag of groceries, washing your scalp, pushing up on your hands, driving etc.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale | 1-2 months
  A total PCS score of 30 represents clinically relevant level of catastrophizing. A total PCS score of 30 corresponds to the 75th percentile of the distribution of PCS scores in clinic samples of chronic pain patients.
Fear Avoidance Beliefs | 1-2 months
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a patient reported questionnaire which measures a patient's fear avoidance beliefs about physical activity and work due to pain and resulting disability
Pain Self-efficacy | 1-2 months
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire, developed to assess the confidence people with ongoing pain have in performing activities while in pain.
Yellow Flag Risk | 1-2 months
  A 17 question questionnaire that predicts and screens risk of pain disability and factors preventing recovery. Patterns suggest pain mechanism; Measures functional outcome from low, moderate, or high risk groups

CONTACTS AND LOCATIONS:
Overall Officials: James Petros, MD, Principal Investigator — Chief Medical Officer
Locations (1):
- Allied Pain & Spine Institute, Los Gatos, California, United States

IPD SHARING:
Plan to Share IPD: No